CLINICAL TRIAL: NCT00669188
Title: Patient-Provider Communication and Interaction in a Virtual Clinical Setting
Brief Title: Patient Provider Communication and Interaction in a Virtual Clinical Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 080122; 08-HG-0122
Record Dates: First submitted 2008-04-29; First posted 2008-04-30 (Estimated); Last update posted 2024-08-12 (Actual); Status verified 2024-01-09

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Information Type 1 (Experimental): genetic risk information
  Interventions: Other: Information
- Information Type 2 (Sham Comparator): information absent
  Interventions: Other: Information absent

INTERVENTIONS:
Other: Information absent — Information
  Arms: Information Type 2
Other: Information — Information
  Arms: Information Type 1

SUMMARY:
Summary:

A few studies have explored factors which influence patient-provider communication in a controlled setting. However, more information is needed about how different factors affect communication so that it can be improved.

Third- and fourth-year medical students may be eligible for this study. Participants are recruited from the Washington, D.C. area.

At the research center, participants will use a virtual reality headset to view a virtual clinic environment and interact with a virtual patient.

After interacting with the virtual patient, participants will complete a questionnaire about their experience within the virtual clinic and other research-related information.

The total time for the study visit is 60 minutes.

Eligibility:

Third- and fourth-year medical students at least 18 years of age. You may not take part in the study if you have a history of seizures and/or are pregnant.

DETAILED DESCRIPTION:
This study will investigate research questions regarding factors influencing patient-provider communication. Participants will interact with a virtual patient in a virtual clinical setting.

Third- or fourth-year medical students may be eligible for this study. Participants are recruited from the Washington, D.C. area.

Study participants will perform one task and complete one set of questions at the study appointment. The task involves viewing a virtual patient s health information and interacting with the virtual patient in a virtual environment clinical scenario. While in the virtual environment, the subject wears a head-mounted video unit that allows him or her to see elements of the environment. The activities in the virtual environment take about 15 minutes. The total time for the study is about 60 minutes.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy adult volunteers who are third or fourth-year medical students. Both men and women over age 18 will be eligible for this study (though in practice the age range is likely to naturally be constrained by the typical age of medical students).

EXCLUSION CRITERIA: 1) persons with seizure or vestibular disorders; 2) women with known pregnancy; 3) persons who are highly prone to motion sickness; 4) those with low, uncorrected vision or hearing; 5) all current and past employees and contractors of

NHGRI; and 6) persons who have received information about the study purpose or procedure from a past participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2008-04-24 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
treatment recommendations | at time of study
  recommendations made for the virtual patient's treatment

CONTACTS AND LOCATIONS:
Overall Officials: Susan Persky, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-HG-0122.html